CLINICAL TRIAL: NCT02580318
Title: Manipulation of Breath Alcohol Tests: Can Specific Techniques Alter Blood Alcohol Concentration Readings?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Luke's Hospital and Health Network, Pennsylvania (Other)
Responsible Party: Principal Investigator, Holly Stankewicz, D.O., Attending physician and faculty emergency medicine resiency, St. Luke's Hospital and Health Network, Pennsylvania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SLHN 2015-28
Record Dates: First submitted 2015-09-10; First posted 2015-10-20 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Alcohol Concentration Values; Alcohol Intoxication
MeSH Terms: conditions — Alcoholic Intoxication | interventions — Breath Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all study participants (Experimental): subjects consumed alcohol to a BrAC of 0.1 and then performed the following manipulations while using the breathalyzer: poor effort, hyperventilation (immediate), hyperventilation (after 5 minutes), hyperventilation (after 10 minutes), drinking water (immediate), drinking water (after 5 minutes)
  Interventions: Device: breathalyzer

INTERVENTIONS:
Device: breathalyzer

SUMMARY:
This is a prospective cohort study. The investigators will enroll 50 healthy volunteers. In a safe environment and after signing informed consent, each participant will consume a standardized alcoholic beverage. Using a Breathalyzer, the subjects BAT will be measured. If the subject's BAT is less than 0.10 +/- 0.005, the subject will drink another alcoholic beverage. This process will continue until the subject's BAT is 0.10 +/- 0.005. The number of alcoholic beverages the subject consumes will be monitored by the observers. When the target BAT is reached, the subjects will manipulate the breathalyzer in various ways and measure their BAT again after each manipulation. In a set order, the subjects will manipulate the breathalyzer by using less than the subject's maximal exhalation effort, placing the breathalyzer at the side of the subject's mouth, hyperventilating (10 rapidly (less than 1 second) and successive breaths prior to using the device), repeating breathalyzer 5 minutes and 10 minutes after hyperventilation and then drinking cold water after the breathalyzer at 10 minutes and repeating the breathalyzer after drinking some cold water. Descriptive statistical analyses as well as Pearson's product moment correlation coefficient will be employed to determine if any statistically significant correlation exists for any of the manipulations.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers over age 21

Exclusion Criteria:

* pregnancy
* alcoholism
* diabetes
* kidney/bladder stones
* kidney disease
* liver disease
* stomach ulcer
* organ transplant patients
* dialysis patients
* subjects with alcohol allergies
* subjects taking the following medications: activated charcoal, ampicillin, carbamazepine, cephaloridine, cloxacillin, methicillin, nitroglycerine, oxacillin, penicillin G, or quinicillin

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Stankewicz, D.O., Principal Investigator — St. Luke's University Hospital
Locations (1):
- St. Luke's Hospital, Bethlehem, Pennsylvania, United States

REFERENCES:
- [Result] Jones AW. Quantitative measurements of the alcohol concentration and the temperature of breath during a prolonged exhalation. Acta Physiol Scand. 1982 Mar;114(3):407-12. doi: 10.1111/j.1748-1716.1982.tb07002.x. PMID 7136772

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 54 participants.
Groups:
- All Study Participants: participants drank beer to a BrAC level of 0.1 and then were instructed to do the following manipulations: poor effort, hyperventilation(immediate), hyperventilation (after 5 minutes), hyperventilation (after 10 minutes), drinking water (immediate), drinking water (after 5 minutes)
Period: Overall Study
Arm/Group | All Study Participants
Started | 54
Poor Effort | 53
Hyperventilation (Immediate) | 54
Hyperventilation (5 Minutes) | 54
Hyperventilation (10 Minutes) | 54
Drinking Water (Immediate) | 51
Drinking Water (5 Minutes) | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Percent Alcohol Concentration Measured by Breathalyzer
Time Frame: 20 minutes
Population: number of participants that completed breath alcohol content are reported.
Measure: Mean (Standard Deviation); unit: percent Breathalyzed alcohol content
Arm/Group | All Study Participants
Number analyzed (Participants) | 54
percent Breathalyzed alcohol content
  poor effort: number analyzed (Participants) | 53
  poor effort | 0.099 (.010)
  hyperventilation (immediate) | 0.086 (0.011)
  hyperventilation (5 minutes) | 0.099 (0.009)
  hyperventilation (10minutes) | 0.099 (0.011)
  drinking water(immediate): number analyzed (Participants) | 51
  drinking water(immediate) | 0.084 (0.011)
  drinking water (5 minutes) | 0.096 (0.013)
Statistical Analysis 1: Comparison: All Study Participants; this p value is calculated for poor effort; Test type: Other; p < 0.0001, t-test, 2 sided — the separate paired sample t-tests were conducted to compare the baseline BrAC to the BrAC after the manipulation (poor effort)
Statistical Analysis 2: Comparison: All Study Participants; p value calculated for hyperventilation (immediate); Test type: Other; p < 0.0001, t-test, 2 sided — the separate paired sample t-tests were conducted to compare the baseline BrAC to the BrAC after the manipulation (hyperventilation - immediate)
Statistical Analysis 3: Comparison: All Study Participants; p value calculated for hyperventilation (after 5 minutes); Test type: Other; p < 0.0001, t-test, 2 sided — the separate paired sample t-tests were conducted to compare the baseline BrAC to the BrAC after the manipulation (5 minutes after hyperventilation)
Statistical Analysis 4: Comparison: All Study Participants; p value calculated for hyperventilation (after 10 minutes); Test type: Other; p < 0.0001, t-test, 2 sided — the separate paired sample t-tests were conducted to compare the baseline BrAC to the BrAC after the manipulation (10 minutes after hyperventilation)
Statistical Analysis 5: Comparison: All Study Participants; p value calculated for drinking water (immediate); Test type: Other; p < 0.0001, t-test, 2 sided — the separate paired sample t-tests were conducted to compare the baseline BrAC to the BrAC after the manipulation (immediately after drinking water)
Statistical Analysis 6: Comparison: All Study Participants; p value calculated for drinking water (5 minutes); Test type: Other; p < 0.0001, t-test, 2 sided — the separate paired sample t-tests were conducted to compare the baseline BrAC to the BrAC after the manipulation (5 minutes after drinking water)

ADVERSE EVENTS:
Time Frame: 12 hours
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 4/54
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=54)
vomiting (Gastrointestinal disorders) | 2
vertigo (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes